CLINICAL TRIAL: NCT01855295
Title: Protein Supplementation in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Srinvasan Beddhu, MD, Professor of Medicine, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00036763
Record Dates: First submitted 2013-04-18; First posted 2013-05-16 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Disease
Keywords: Dialysis; End Stage Renal Disease; Protein supplementation; Inflammation; Quality of Life
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Protein Supplementation (Experimental): Hemodialysis patients with inflammation and low body mas index to receive protein dietary advice and protein supplements while on dialysis
  Interventions: Dietary Supplement: Protein Supplement

INTERVENTIONS:
Dietary Supplement: Protein Supplement — During the treatment phase, study subjects are advised to increase protein intake to 1.2 g/kg/day for 12 weeks. In addition to any protein supplementation the participant is on, supervised supplementation on each dialysis session is provided. Each participant receives 45 grams of liquid protein supplement (Provide Sugar Free produced by Provide Nutrition LC) at each dialysis treatment for additional 12 weeks for total study duration of 24 weeks.

SUMMARY:
Poor nutritional status as evidenced by low body mass index, low muscle mass or low serum albumin is a strong predictor of morbidity and mortality in dialysis patients. Hypercatabolism induced by inflammation is widely considered the cause of uremic malnutrition even though there is no clear evidence that hemodialysis patients with elevated C-reactive protein (CRP) levels are at greater risk of losing weight or muscle mass. Conversely, there is little data on whether dialysis patients with malnutrition and elevated C-reactive protein levels would gain muscle mass with protein supplementation.

The hypothesis is that protein supplementation during dialysis will improve muscle mass, functional status and quality of life in inflamed malnourished hemodialysis patients. Therefore, the objectives of the current proposal are to examine in malnourished (body mass index < 23 kg/m2 or serum creatinine < 8 mg/dL) hemodialysis patients with inflammation (high sensitivity CRP > 3 mg/dL), the effects of protein supplementation on

1. Muscle mass as determined by creatinine kinetics
2. Functional status as assessed by 6 min walk
3. Quality of life as assessed by Short Form -12 survey

DETAILED DESCRIPTION:
Design: Open labeled trial.

Recruitment and Randomization: Men and women aged 18 or older receiving care at the University of Utah dialysis centers.

Study procedures: Men and women on hemodialysis for at least for 3 months with malnutrition (defined as Body Mass Index less than 23 kg/m2 or serum creatinine < 8 mg/dL) will be approached to determine whether they want to participate in the study. If they are interested, the study purpose and procedures will be explained and informed consent obtained. 5 ml of screening blood will be obtained before dialysis to measure CRP. If it is greater than > 3 mg/dL, that individual will be eligible to participate in the study. Participants will be asked to complete a brief questionnaire on demographics (age, gender, race, education), comorbid conditions, physical activity level and quality of life. Height, weight, and waist circumference will be measured. Relevant data on dialysis, medications, laboratory markers will be obtained from the electronic medical records.

The investigators anticipate to obtain screening blood draw in about 80 participants and that about half of these will have elevated CRP and qualify to participate in the study. The 40 participants will receive dietary advice to increase protein intake to 1.2 g/kg/day and monitored for 12 weeks. Then, each participant will receive 45 grams of liquid protein supplement at each dialysis treatment for additional 12 weeks for total study duration of 24 weeks. Compliance and tolerance of the supplement will be monitored.

Protein supplementation such as Boost, Procel or liquid supplements is used regularly in dialysis patients. The protein supplement used in the study is Provide Sugar Free produced by Provide Nutrition LC. The Food and Drug Administration regulates it as a nutrition supplement. It is a liquid supplement made from enzyme hydrolyzed collagen protein. This supplement is used in malnutrition, bariatric surgery, dialysis, poor appetite, and wound care. The investigators chose this supplement because the investigators were able to get it at a reduced cost. There is no data available to show that this supplement is better or worse than any other supplements currently available. The manufacturer states that the sugar free Provide is phosphorous free. However, the investigators will monitor phosphorous levels in the study patients.

Pre-dialysis blood sample (15 ml in lithium heparin tube) and post dialysis blood sample (5 ml in lithium heparin tube) will be drawn at baseline, 4, 12, 16 and 20 weeks. Pre and post dialysis creatinine along with 44-hour urine collection for creatinine will be obtained at baseline 4, 12, 16 and 24 weeks for estimating muscle mass using creatinine kinetics. Short Form -12 survey for quality of life will be obtained at baseline 4, 12, 16, and 24 weeks. Distances walked during in 6-minutes will be recorded at baseline, 4, 12, 16 and 24 weeks.

Assays of Serum analytes:

1. Interleukin-6 (IL-6): The measurement of serum IL-6 will be performed using an IMMULITE 1000 analyzer and reagents from Diagnostic Products Corporation. The performance characteristics of this immunoassay include an analytic measurement range of 2 to 1000 pg/mL, imprecision of <7.6% from 88 to 1000 pg/mL, and a reference interval of <6 pg/mL.
2. Tumor necrosis factor-alpha (TNF-alpha): The measurement of serum TNF- alpha will be performed using an IMMULITE 1000 analyzer and reagents from Diagnostic Products Corporation. The performance characteristics of this immunoassay include an analytic measurement range of 2 to 1000 pg/mL, imprecision of <6.6% from 17 to 788 pg/mL, and a reference interval of <8 pg/mL.
3. high sensitivity CRP: The measurement of serum C-reactive protein will be performed using the FDA-cleared Roche Tina-quant latex high sensitivity kit on a Roche MODULAR P analyzer. The performance characteristics of this turbidimetric assay include an analytic measurement range of 0.1 to 20 mg/L and imprecision of <5.8%.
4. Insulin: The measure of insulin will be performed using a Diagnostic Products Corporation kit on an IMMULITE 2000 analyzer. The performance characteristics of this immunoassay include an analytic measurement range of 2 to 300 mIU/L , imprecision of <7.4% from 8 to 291 mIU/L, and a fasting reference interval of <29 mIU/L.

ELIGIBILITY:
Inclusion criteria

* Subjects (men and women) on hemodialysis for at least 3 months
* Inflammation (high sensitivity CRP > 3 mg/dL)
* Body Mass Index < 23 kg/m2; or low muscle mass as evidenced by serum creatinine < 8 mg/dL in the presence of anuria (urine output < 200 ml/d) and adequate dialysis (Urea Reduction Ratio > 65%).

Exclusion criteria

* Pregnant subjects
* Subjects who are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Protein Stores as measured by mid arm circumference (cm) | Baseline to 24 weeks
  Triceps skin fold thickness and mid-arm muscle arm circumference are measured to assess protein stores.